CLINICAL TRIAL: NCT01277965
Title: Use of a CMGS to Validate Algorithms for Basal Insulin Rate Reductions in Type 1 Diabetic Patients Treated With Subcutaneous Continuous Insulin Infusion and Practicing Physical Activity
Brief Title: Validation of Algorithms for Basal Insulin Rate Reductions in Type 1 Diabetic Patients Practising Physical Activity
Acronym: DIABRASPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: European Association for the Study of Diabetes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2009 A01136 51
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2012-01

CONDITIONS: Type 1 Diabetes With a Subcutaneous Insulin Pump; Adjustment of the Recommended Basal Insulin Flow Rate in the Event of Physical Activity; Adjustment of the Recommended Prandial Insulin in the Event of Physical Activity
Keywords: Algorithm basal insulin; physical activity; Type 1 diabetes; Insulin pump treatment
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 1 | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 50% VO2 max, BFR reduced by 50% (Other): The basal rate of the pump will be adjusted in accordance with the intensity of physical activity being performed for moderate physical activity (50% VO2max),a temporary basal rate will be reduced by 50%
  Interventions: Other: 50%VO2maxTBR50
- 50% VO2 max,BFR reduced by 80% (Other): The basal rate of the pump will be adjusted in accordance with the intensity of physical activity being performed for moderate physical activity (50% VO2max),a temporary basal rate will be reduced by 80%
  Interventions: Other: 50%VO2max TBR80
- 75% VO2 max, BFR reduced by 80% (Other): The basal rate of the pump will be adjusted in accordance with the intensity of physical activity being performed for moderate physical activity (75% VO2max),a temporary basal rate will be reduced by 80%.
  Interventions: Other: 75%VO2max TBR80
- 75% VO2 max, pump switched off (Other): Turning off the pump (75%VO2max TBR100).However, in order to maintain the study blindfold, the pump will be switched off but not removed.
  Interventions: Other: 75%VO2max TBR100
- Rest (Other): Patient will be in rest, basal insulin flow rate will not be change.
  Interventions: Other: Rest

INTERVENTIONS:
Other: 50%VO2maxTBR50 — The basal rate of the pump will be adjusted in accordance with the intensity of physical activity being performed for moderate physical activity (50% VO2max),a temporary basal rate will be reduced by 50%
  Arms: 50% VO2 max, BFR reduced by 50%
Other: 50%VO2max TBR80 — The basal rate of the pump will be adjusted in accordance with the intensity of physical activity being performed for moderate physical activity (50% VO2max),a temporary basal rate will be reduced by 80%
  Arms: 50% VO2 max,BFR reduced by 80%
Other: 75%VO2max TBR80 — The basal rate of the pump will be adjusted in accordance with the intensity of physical activity being performed for moderate physical activity (75% VO2max),a temporary basal rate will be reduced by 80%
  Arms: 75% VO2 max, BFR reduced by 80%
Other: 75%VO2max TBR100 — Turning off the pump (75%VO2max TBR100).However, in order to maintain the study blindfold, the pump will be switched off but not removed
  Arms: 75% VO2 max, pump switched off
Other: Rest — Patient will be in rest, basal insulin flow rate will not be change
  Arms: Rest

SUMMARY:
Primary aim:

To show that in subjects with type 1 diabetes with a subcutaneous continuous insulin infusion, adjustment of the recommended basal insulin flow rate in the event of physical activity allows the subjects to practice sports without any increase in incidence of hypoglycaemia during physical activity or the ensuing hours.

(NB: hypoglycaemia is defined as blood glucose less than 3 mmol/l or 0,54 g/l in accordance with the EMEA definition).

The proposed algorithms consist of a temporary reduction in basal flow of 50 percent or 80 percent (temporary basal flow TBR50 or TBR80) depending on the intensity of physical activity (50 percent of VO2max or 75 percent of VO2max). Switching off the pump will also be studied as an option to adjust insulin dosage in the event of unprogrammed physical activity (temporary reduction of basal flow by 100 percent).

Secondary aims:

* Characterisation of hypoglycaemia during and after physical activity based on CGMS data: symptomatic or non-symptomatic nature of hypoglycaemia, time to onset of hypoglycaemia in relation to the start of physical activity, degree and severity of hypoglycaemia.
* Evaluation of overall variations in blood glucose in the event of physical activity using CGMS data (area under the curve).
* Evaluation of glucose restoration methods used in the event of hypoglycaemia.
* Analysis of subgroups of patients with and without hypoglycaemia.

DETAILED DESCRIPTION:
Inclusion criteria:

* Patients aged over 18 years, presenting type 1 diabetes for at least 1 year
* Patients on basal-prandial regimen treated with functional insulin therapy
* Patients with a subcutaneous insulin pump for at least 3 months
* Patients with HbA1c less than 9 percent less than 3 months before
* Patients with stable basal flow for at least 1 week
* Patients able to pedal
* Patients covered by social security
* Patients consenting to take part in the study and having signed a written informed consent form.

Non-inclusion criteria:

* Patients with a history of severe hypoglycaemia in the 6 months prior to entry into the study
* Patients unable to detect their hypoglycaemia
* Patients with perforating foot ulcer or a known history of heart disease or obliterative arteriopathy of the lower limbs, or a history of cerebrovascular accident, or ongoing proliferative retinopathy or renal failure.
* Patients with poorly controlled hypertension
* Women either pregnant or likely to become pregnant
* Patients deprived of liberty by judicial or administrative decision, patients placed under legal guardianship.

Primary criterion:

Number of episodes of symptomatic or non-symptomatic hypoglycaemia detected by CGMS throughout the duration of physical activity and subsequent hours until the next morning (threshold: 3 mmol/l or 0,54 g/l).

Secondary criteria:

Duration of hypoglycaemia (min), total time in hypoglycaemia (min, percent), time to onset of hypoglycaemia after the start of physical activity, degree (blood glucose level) and severity of hypoglycaemia, area under the algebraic curve during physical activity and in the following hours, nadir of the intervening glucose curve.

Before starting this study, patients will undergo effort testing and measurement of their VO2max in order to precisely define the different thresholds of physical activity.

Tests and proposed insulin adjustment:

- Tests: Basal period

Each patient will undergo 5 consecutive tests over a 6-month period. The tests will be performed 3 hours after the start of the midday meal in order to define a period during which blood glucose is solely dependent on basal flow. The 5 tests will comprise 4 physical tests and 1 resting test, to be performed in random order:

* The 4 physical tests will comprise 2 different levels of intensity (50 percent VO2max, 75 percent VO2max). At each of these levels, patients will test 2 insulin dose adjustment algorithms concerning only the basal flow rate of the insulin pump:
* 50 percent VO2max, TBR reduced by 50 percent (50 percent VO2maxTBR50),
* 50 percent VO2max, TBR reduced by 80 percent (50 eprcent VO2max TBR80)
* 75 percent VO2max, TBR reduced by 80 percent (75 percent VO2max TBR80)
* 75 percent VO2max, pump switched off (75 percent VO2maxTBR100)
* A resting test will be used as a comparator.

Each physical test will comprise testing on a bicycle ergometer for 40 minutes with:

* a 5-minute period during which the intensity of physical activity will be raised
* a 30-minute plateau at the desired intensity and power
* a 5-minute recovery period. "Prandial" period In the second phase, two further tests at 50 percent VO2max will be performed 90 minutes after the start of the meal in order to evaluate the effect of reducing the rapid-acting insulin bolus at the onset of hypoglycaemia.

At the same time, during the 2 periods ("basal" and "prandial"), patients will be asked to score the intensity of their physical activity on the Borg RPE rating scale.

- Adjustment of insulin dose:

* The bolus for the meal preceding physical activity (lunch) will be given as usual, with no deliberate reduction for the ensuing sport.
* "Basal" period

The adjustments in basal flow proposed at the time of physical activity will take into account the intensity of the ensuing physical activity:

* moderate physical activity (50 percent VO2max)
* intense physical activity (75 percent VO2max) with 2 possible options:
* reduction of basal flow by 50 percent or by 80 percent in the first case
* reduction of basal flow by 80 percent or switching off the pump in the second case.

In the event of reduced basal flow, this will be maintained throughout the duration of physical activity and for the 2 hours following the end of physical activity. If the pump is switched off, it will remain switched off throughout the entire duration of physical activity, but it will not be removed in order to maintain the study blind. It will be switched on again routinely at the end of the physical activity period, at the same flow rate as that set prior to physical activity.

- Continuous Monitoring Glucose System (CMGS)

A CMGS to record intervening blood glucose levels will be fitted before lunch and worn until the next morning. Data recorded by the CMGS will not be visible to patients in order to prevent them from attempting to modify their insulin doses based on these values.

Patients will have dinner at 8 o'clock in the evening in their own home in order to allow superimposition of the blood glucose curves and facilitate their interpretation. The CMGS will be removed the next morning after breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years, presenting type 1 diabetes for at least 1 year
* Patients on basal-prandial regimen treated with functional insulin therapy
* Patients with a subcutaneous insulin pump for at least 3 months
* Patients with HbA1c < 9% less than 3 months before
* Patients with stable basal flow for at least 1 week
* Patients able to pedal
* Patients covered by social security
* Patients consenting to take part in the study and having signed a written informed consent form.

Exclusion Criteria:

* Patients with a history of severe hypoglycaemia in the 6 months prior to entry into the study
* Patients unable to detect their hypoglycaemia
* Patients with perforating foot ulcer or a known history of heart disease or obliterative arteriopathy of the lower limbs, or a history of cerebrovascular accident, or ongoing proliferative retinopathy or renal failure.
* Patients with poorly controlled hypertension
* Women either pregnant or likely to become pregnant
* Patients deprived of liberty by judicial or administrative decision, patients placed under legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of episodes of symptomatic or non-symptomatic hypoglycaemia | 24 hours
  Number of episodes of symptomatic or non-symptomatic hypoglycaemia detected by CGMS throughout the duration of physical activity and subsequent hours until the next morning (threshold: 3 mmol/l or 0.54 g/l).

SECONDARY OUTCOMES:
Duration of hypoglycaemia | 24 hours
  Duration of hypoglycaemia (min), total time in hypoglycaemia (min, %), time to onset of hypoglycaemia after the start of physical activity, degree (blood glucose level) and severity of hypoglycaemia, area under the algebraic curve during physical activity and in the following hours, nadir of the intervening glucose curve.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia FRANC, PH, Principal Investigator — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, Essonne, France